CLINICAL TRIAL: NCT01673022
Title: Determining the Sensitivity of Sentinel Lymph Nodes Identified With Robotic Fluorescence Imaging for Detecting Metastatic Endometrial and Cervical Cancer
Brief Title: Determining the Sensitivity of Sentinel Lymph Nodes Identified With Robotic Fluorescence Imaging
Acronym: FIRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1204008493
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2017-07

CONDITIONS: Endometrial Cancer; Cervical Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — Indocyanine Green; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IC Green Arm (Experimental): One arm only: Receives IC Green for testing of study objective
  Interventions: Drug: IC Green

INTERVENTIONS:
Drug: IC Green — IC Green
  Other Names: indocyanine green for injection, USP

SUMMARY:
Description:

This is a multi-institutional study investigating the sensitivity and negative predictive value of sentinel lymph nodes mapped with robotic assisted near infrared imaging after cervical injection of indocyanine green (ICG) dye for women with stage I endometrial or cervical cancer at the time of their robotic surgical staging.

Patients will receive cervical injection of 1mg ICG after induction of anesthesia followed by sentinel lymph node mapping using robotic assisted fluorescence imaging. The sentinel lymph nodes identified will be removed and sent for ultraprocessing by pathology. The non-sentinel pelvic and para-aortic (if indicated) non-sentinel nodes will be removed and sent for routine pathologic processing according to standard of care for these surgical procedures. The pathologic results of the sentinel and non-sentinel nodes will be evaluated for sensitivity and negative predictive value in their ability to detect metastatic disease.

DETAILED DESCRIPTION:
Brief Summary:

Patients with early stage endometrial and cervical cancer who are undergoing robotic surgery to remove the uterus, cervix and lymph nodes will have dye injected into the cervix after they are asleep from anesthesia prior to performing the surgery. During the surgery, the surgeon will activate the robotic camera that is being used to visualize the internal organs changing it to a special mode of imaging called near infrared imaging. The near infrared imaging will allow the surgeon to see where the dye that was injected into the cervix has spread. The dye travels through vessels called lymphatic channels to nodules called "sentinel lymph nodes". These are the tissues the surgeon is most interested in removing in order to see if there has been spread of their cancer to those nodules. The dye that travels to the lymph nodes makes them more easily visible to the surgeon. Without the dye, these nodes are indistinguishable from the surrounding fatty tissue.

The nodes that have dye in them will be removed from the patient and sent to the pathologist, where they will be very closely examined, called ultrasectioning, for cancer spread. The surgeon will remove the remaining lymphatic tissue (all of the fatty and lymphatic tissue that surrounded the sentinel lymph node that did not stain with the dye), as these are the "non-sentinel lymph nodes", and are the tissue that is traditionally removed with endometrial and cervical cancer surgery as part of standard of care. These non-sentinel lymph nodes will also be examined for evidence of cancer spread. The researchers will compare the pathology results from the sentinel nodes and non-sentinel nodes. The researchers hypothesize that the sentinel nodes contain cancer cells at least 90% of the time when there is cancer found in the non-sentinel nodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be women 18 years and older who have biopsy proven endometrial or cervical carcinoma (of any histologic subtype).
* Surgical staging with the da Vinci Si robotic tool must be planned with a planned pelvic and, in the case of endometrial cancer, a para-aortic lymphadenectomy
* Patients must meet criteria for robotic surgical approach:
* Patients must have either a clinical stage I endometrial (of any histologic grade) or FIGO stage IA2 or IB1 (<4cm) cervical squamous, adenocarcinoma or adenosquamous carcinoma.
* Patients must be able to sign an informed consent in English language.
* Patients with known liver disease will require normal range liver function tests as determined by pre-operative labs drawn within 30 days of surgery.

Exclusion Criteria:

* Patients who have iodide allergies
* Patients who have had previous retroperitoneal surgery
* Patients on whom pelvic+/- para-aortic lymphadenectomy is not planned as part of their surgical staging.
* Patients who have received previous treatment for their endometrial or cervical cancer (particularly hysterectomy or pelvic radiation).
* Patients who are pregnant.
* Patients with documented liver disease who have abnormalities of liver function tests.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2012-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Rossi, MD, Principal Investigator — Indiana University
Locations (7):
- United States (7):
  - USA Mitchell Cancer Institute, Mobile, Alabama
  - Indiana University, Indianapolis, Indiana
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - University of North Carolina, Chapel Hill, North Carolina
  - Tri Health Good Smaritan Hospital, Cincinnati, Ohio
  - University of Virginia Medical Center, Charlottesville, Virginia

REFERENCES:
- [Derived] Rossi EC, Kowalski LD, Scalici J, Cantrell L, Schuler K, Hanna RK, Method M, Ade M, Ivanova A, Boggess JF. A comparison of sentinel lymph node biopsy to lymphadenectomy for endometrial cancer staging (FIRES trial): a multicentre, prospective, cohort study. Lancet Oncol. 2017 Mar;18(3):384-392. doi: 10.1016/S1470-2045(17)30068-2. Epub 2017 Feb 1. PMID 28159465

RESULTS

PARTICIPANT FLOW:
Groups:
- IC-GREEN® (Indocyanine Green) Arm: One arm only: Receives IC-GREEN® (Indocyanine green) for testing of study objective
  IC-GREEN®: Indocyanine green
Period: Overall Study
Arm/Group | IC-GREEN® (Indocyanine Green) Arm
Started | 430
Completed | 422
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | IC Green Arm
Number analyzed (Participants) | 430
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 293
  >=65 years | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 430
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 430

OUTCOME MEASURES:

1. Primary Outcome: Estimate the Sensitivity of the Sentinel Lymph Node
Description: To estimate the sensitivity of the sentinel lymph node in the determination of lymph node metastases in patients with invasive carcinoma of the cervix and uterus using Indocyanine Green (ICG) and robotic assisted near infrared (NIR) imaging. Sensitivity is defined as the proportion of sentinel lymph node: number of participants with, determined to be metastatic by both IGR/NIR and pathology out of the sentinel lymph nodes found to be metastatic by pathology.
Time Frame: 3 years
Population: Sensitivity of the sentinel lymph node
Measure: Count of Participants; unit: Participants
Groups:
- IC Green (Indocyanine Green) Arm: One arm only: Receives IC Green (indocyanine green) )for testing of study objective
  IC Green: IC Green (indocyanine green)
Arm/Group | IC Green (Indocyanine Green) Arm
Number analyzed (Participants) | 430
Participants | 418

ADVERSE EVENTS:
Arm/Group | IC Green Arm
Serious Adverse Events (participants affected / at risk) | 22/430
Other Adverse Events (participants affected / at risk) | 17/430
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IC Green Arm (N=430)
postoperative respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4
postoperative neurological disorder (Nervous system disorders) | 4
ureteral injury (Renal and urinary disorders) | 1
nausea (Gastrointestinal disorders) | 5
pain (Surgical and medical procedures) | 4
anemia (Blood and lymphatic system disorders) | 1
syncope (Cardiac disorders) | 1
lymphedema (Skin and subcutaneous tissue disorders) | 1
hemorrhage (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IC Green Arm (N=430)
abdominal pain (Surgical and medical procedures) | 3
hypokalemia (Blood and lymphatic system disorders) | 2
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
hypertension (Cardiac disorders) | 1
hypotension (Cardiac disorders) | 2
dizziness (Nervous system disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 1
fever (Infections and infestations) | 3
anemia (Blood and lymphatic system disorders) | 2
nausea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No